CLINICAL TRIAL: NCT05648916
Title: The Effect of Celecoxib on Heterotopic Bone Formation Following Cementless Total Hip Arthroplasty
Brief Title: Celebrex and HO Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Adam Hart, Staff Orthopaedic Surgeon, Clinical Researcher, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2023-8872
Record Dates: First submitted 2022-11-23; First posted 2022-12-13 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Heterotopic Ossification
Keywords: heterotopic ossification; celecoxib; arthroplasty
MeSH Terms: conditions — Ossification, Heterotopic | interventions — Celecoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with and without HO before Celecoxib clinical pathway: Patients with and without heterotopic ossification (HO) before the clinical pathway was changed to include celecoxib following cementless total hip joint replacement surgery between periods 2009-2012.
- Patients with and without HO after Celecoxib clinical pathway: Patients with and without heterotopic ossification (HO) after the clinical pathway was changed to include celecoxib following cementless total hip joint replacement surgery between periods 2013-2020.
  Interventions: Other: Celecoxib

INTERVENTIONS:
Other: Celecoxib — Retrospectively comparing patients with and without heterotopic ossification who have been exposed to celecoxib and underwent cementless total hip joint replacement surgery.
  Other Names: Celebrex
  Groups: Patients with and without HO after Celecoxib clinical pathway

SUMMARY:
The primary goal of this observational study is to demonstrate the incidence of heterotopic ossification (HO) in patients with cementless total hip joint replacement surgery over time and secondly, demonstrate the relationship between celecoxib and HO formation. Lastly, investigators will examine the relationship between HO and patient-reported outcome measures (PROMs).

DETAILED DESCRIPTION:
Heterotopic ossification (HO) is characterized by the pathologic formation of mature lamellar bone in muscle and soft tissue. It presents clinically with localized pain, reduced motion, and swelling. The process of HO occurs due to abnormal tissue repair, and most commonly occurs in young adults. Significant predisposing factors include total hip arthroplasty (THA), fractures, spinal cord and traumatic brain injuries, and thermal injuries. The overall incidence of HO is up 42% to 57% after THA, and the incidence of extensive HO post THA is 2% to 7%. Certain patient and surgical-related factors have been associated with an increased risk of HO. Patient aspects include a history of Paget's disease, ankylosing spondylitis, and hypertrophic osteoarthritis; surgical factors include the use of cemented implants and prolonged time of ischemia. Post-operative celecoxib use has been associated with a significant lower incidence of HO compared to controls. Furthermore, among COX-2 selective inhibitors, celecoxib has been associated with the lowest incidence of HO.

This study looks at patients who have been referred to our orthopaedic clinic and undergone cementless total hip joint replacement surgery through a retrospective review of our pre-existing departmental database. All the data from all patients who meet the inclusion criteria will be collected from our database. Specifically, the age, gender, BMI, pre-operative diagnosis, post operative radiotherapy, preoperative patient-reported outcome measures (PROMs), post-operative PROMs, operative characteristics, and complications. Data from the available PROMs database will need to be converted into a manageable format that is suitable for data analysis. This study looks at the Harris Hip Score, the UCLA Activity Score, and SF-12 PROMs that are collected from each patient as standard of care. Descriptive statistics and para/nonparametric statistics will be used to analyze the data through IBM SPSS software platform for statistical analysis. The independent student t-test and multivariable logistic regression analysis will be used to examine outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* All primary total hip replacements with Cementless Tri-lock BPS (Depuy, Warsaw, IN) with minimum 2 years follow up.

Exclusion Criteria:

* Revision surgery
* Infections
* Other implants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been referred to our outpatient orthopaedic clinic and undergone cementless total hip joint replacement surgery.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of heterotopic ossification (HO) in patients with cementless total hip joint replacements over time. | 10 mins
  The percentage of patients with HO who have undergone cementless total hip joint replacement surgery over time.

SECONDARY OUTCOMES:
The association between celecoxib and patients with and without heterotopic ossification (HO) following cementless total hip joint replacements. | 10 mins
  The probability between the use of celecoxib and patients with and without heterotopic ossification following cementless total hip joint replacement surgery.
The association between heterotopic ossification (HO) and celecoxib and between HO and patient-reported outcome measures in patients with cementless total hip joint replacements. | 10 mins
  The probability between heterotopic ossification (HO) and the use of celecoxib and between HO and patient-reported outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Hart, MD, Principal Investigator — Research Institute of the McGill University Health Centre
Locations (1):
- Dr, Adam Hart, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhu Y, Zhang F, Chen W, Zhang Q, Liu S, Zhang Y. Incidence and risk factors for heterotopic ossification after total hip arthroplasty: a meta-analysis. Arch Orthop Trauma Surg. 2015 Sep;135(9):1307-14. doi: 10.1007/s00402-015-2277-8. Epub 2015 Jul 9. PMID 26155968
- [Background] Meyers C, Lisiecki J, Miller S, Levin A, Fayad L, Ding C, Sono T, McCarthy E, Levi B, James AW. Heterotopic Ossification: A Comprehensive Review. JBMR Plus. 2019 Feb 27;3(4):e10172. doi: 10.1002/jbm4.10172. eCollection 2019 Apr. PMID 31044187
- [Background] Pai VS. Heterotopic ossification in total hip arthroplasty. The influence of the approach. J Arthroplasty. 1994 Apr;9(2):199-202. doi: 10.1016/0883-5403(94)90069-8. PMID 8014651
- [Background] Gebuhr P, Sletgard J, Dalsgard J, Soelberg M, Keisu K, Hanninen A, Crawford M. Heterotopic ossification after hip arthroplasty: a randomized double-blind multicenter study tenoxicam in 147 hips. Acta Orthop Scand. 1996 Feb;67(1):29-32. doi: 10.3109/17453679608995604. PMID 8615097
- [Background] Riegler HF, Harris CM. Heterotopic bone formation after total hip arthroplasty. Clin Orthop Relat Res. 1976 Jun;(117):209-16. PMID 1277668
- [Background] Ritter MA, Sieber JM. Prophylactic indomethacin for the prevention of heterotopic bone formation following total hip arthroplasty. Clin Orthop Relat Res. 1985 Jun;(196):217-25. PMID 3995821
- [Background] Joice M, Vasileiadis GI, Amanatullah DF. Non-steroidal anti-inflammatory drugs for heterotopic ossification prophylaxis after total hip arthroplasty: a systematic review and meta-analysis. Bone Joint J. 2018 Jul;100-B(7):915-922. doi: 10.1302/0301-620X.100B7.BJJ-2017-1467.R1. PMID 29954195
- [Background] Oni JK, Pinero JR, Saltzman BM, Jaffe FF. Effect of a selective COX-2 inhibitor, celecoxib, on heterotopic ossification after total hip arthroplasty: a case-controlled study. Hip Int. 2014 May-Jun;24(3):256-62. doi: 10.5301/hipint.5000109. Epub 2014 Jan 28. PMID 24474408
- [Background] Saudan M, Saudan P, Perneger T, Riand N, Keller A, Hoffmeyer P. Celecoxib versus ibuprofen in the prevention of heterotopic ossification following total hip replacement: a prospective randomised trial. J Bone Joint Surg Br. 2007 Feb;89(2):155-9. doi: 10.1302/0301-620X.89B2.17747. PMID 17322426
- [Background] Haffer H, Muller M, Ascherl R, Perka C, Winkler T. Diclofenac for prophylaxis of heterotopic ossification after hip arthroplasty: a systematic review. Hip Int. 2022 Mar;32(2):144-151. doi: 10.1177/1120700020978194. Epub 2020 Dec 3. PMID 33272062
- [Background] Harris WH. Traumatic arthritis of the hip after dislocation and acetabular fractures: treatment by mold arthroplasty. An end-result study using a new method of result evaluation. J Bone Joint Surg Am. 1969 Jun;51(4):737-55. No abstract available. PMID 5783851
- [Background] Zahiri CA, Schmalzried TP, Szuszczewicz ES, Amstutz HC. Assessing activity in joint replacement patients. J Arthroplasty. 1998 Dec;13(8):890-5. doi: 10.1016/s0883-5403(98)90195-4. PMID 9880181
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Brooker AF, Bowerman JW, Robinson RA, Riley LH Jr. Ectopic ossification following total hip replacement. Incidence and a method of classification. J Bone Joint Surg Am. 1973 Dec;55(8):1629-32. No abstract available. PMID 4217797